CLINICAL TRIAL: NCT06023238
Title: Antibiotic Elution Profile and Outcomes in the Treatment of Prosthetic Joint Infections of the Knee
Brief Title: Knee Prosthetic Joint Infection Antibiotic Elution
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, F. Johannes Plate, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY22070087
Record Dates: First submitted 2023-08-14; First posted 2023-09-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prosthetic-joint Infection; Arthroplasty Complications
Keywords: Prosthetic Joint Infection; Revision Total Knee Arthroplasty; Antibiotic Elution Profile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid obtained in the post-operative setting as part of standard of care intra-articular post-operative drains or as part of standard of care intra-articular knee aspiration performed during re-implantation revaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic TKA PJI Group: Patients presenting for surgical management of a chronic total knee arthroplasty (TKA) prosthetic joint infection (PJI). Patients will be excluded if they are less than 18 years of age, have a prior history of ipsilateral or contralateral PJI warranting operative management, or are unable to provide informed consent.
  Interventions: Procedure: Treatment of Chronic TKA PJI

INTERVENTIONS:
Procedure: Treatment of Chronic TKA PJI — Patients will all undergo standard of care treatment for a chronic total knee arthroplasty prosthetic joint infection.

SUMMARY:
Patients presenting with prosthetic joint infections of a total knee replacement who are treated with an antibiotic spacer will be observed prospectively for their response to treatment and antibiotic elution profiles will be measured post-operatively utilizing mass spectrometry from synovial fluid acquired as part of standard of care in the management of prosthetic joint infection. Secondary outcomes including post-operative complications, re-operation rates, and re-admission rates will also be compared.

DETAILED DESCRIPTION:
The current study aims to assess the surgical and patient-reported outcomes and in vivo antibiotic elution profile of the management of total knee arthroplasty (TKA) prosthetic joint infection (PJI). Within the standard of care, TKA PJI is treated via a resection arthroplasty and antibiotic cement spacer placement. Patients will be enrolled if they are undergoing surgical management for a chronic TKA PJI and will receive surgical treatment according to the standard of care. In the post-operative period, patients will be monitored for surgical and patient-reported outcomes including re-operation rate, pain scores, complication rates, and re-infection rates. Synovial fluid obtained from intra-articular postoperative drains and at postoperative knee aspirations during reimplantation evaluations will also be utilized for antibiotic concentration quantification via mass spectrometry, if sufficient specimen is available. Patient who undergo surgical management for their chronic TKA PJI will then have their measured antibiotic elution concentrations compared. The study hypothesizes that patients undergoing treatment of a PJI with antibiotic spacer + antibiotic cement spacer will have better surgical and patient-related outcomes with higher antibiotic elution concentrations. These improved outcomes would include lower re-operation rates, lower pain scores, lower wound healing complications, and higher rates of second stage re-implantation observed in patients with higher antibiotic elution concentrations.

Specific aims:

1. To evaluate the antibiotic elution profile and post-operative intra-synovial concentrations in the treatment of chronic PJI after TKA.
2. To evaluate surgical and patient-related outcomes in chronic TKA PJI patients following implant resection and knee spacer placement, including amount of post-operative drain output, wound healing complications, 30- and 90-day risk of re-operation, pain scores, and rate of second stage re-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for treatment of a total knee arthroplasty prosthetic joint infection
* Patients greater than 18 years of age
* Patients able to provide informed consent

Exclusion Criteria:

* Prior history of ipsilateral or contralateral prosthetic joint infection warranting operative management
* Patients less than 18 years of age
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of patients who have had a previous total knee arthroplasty (TKA), presenting with clinical and laboratory findings concerning for a chronic TKA prosthetic joint infection (PJI) undergoing staged surgical management consisting of resection arthroplasty followed by mobile antibiotic spacer placement. Patients who have had prior surgical treatment of a PJI and are less than 18 years of age will not be included in the study population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Intra-articular Antibiotic Elution Profile | Post-operative day 2 and during 2nd stage re-implantation evaluation (around 10 weeks according to standard of care)
  Antibiotic concentration will be quantified utilizing mass spectrometry from intra-articular synovial fluid obtained from post-operative drain and knee aspirations performed for re-implantation evaluation.

SECONDARY OUTCOMES:
Drain Output | Each 12 hours period until removal of the drain up to 5 days postoperatively based on drain output less than 30cc in 12 hours.
  Measured volume of output from post-operative drain will be quantified every 12 hours
Wound Healing Complications | up to 6 months following surgery
  Any issues with wound healing including closure, occurrence of infection, high drainage, or hematoma formation will be among wound healing complications which are measured.
Re-operation Rates | 30 days and 90 days post-operatively.
  Rates of return to operating room will be quantified over course of 30 days and 90 days.
Re-admission Rates | 30 days and 90 days post-operatively.
  Rates of re-admission will be quantified over course of 30 days and 90 days.
Pain Scores | Daily on postop day 0 until postop day 5, 3 weeks, 6 weeks and 10 weeks, 6 months postoperatively.
  Pain scores utilizing visual analog scale from 0 to 10 will be quantified during post-operative course.
Second Stage Re-implantation Rates | Through study completion up to 1 year
  Rates of successful second stage re-implantation will be quantified during the post-operative course.
Knee aspiration cell count | 3 weeks, 6 weeks and 10 weeks - 6 months postoperatively.
  Knee aspiration with number of white cells less than 1300
Knee aspiration culture | 3 weeks, 6 weeks and 10 weeks - 6 months postoperatively.
  Knee aspiration without evidence of bacteria on bacterial culture
C-reactive protein assessment | baseline, 10 weeks to 6 months posteroperatively
  C-reactive protein normalization (less than 1mg/dl)
ESR assessment | baseline, 10 weeks to 6 months posteroperatively
  Erythrocyte sedimentation rate normalization (less than 20 mm/hr)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes F Plate, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
There are no plans at present to make individual participant data (IPD) available to other researchers, however we may share de-identified data with other researchers in the future.

REFERENCES:
- [Background] Chen AF, Parvizi J. Antibiotic-loaded bone cement and periprosthetic joint infection. J Long Term Eff Med Implants. 2014;24(2-3):89-97. doi: 10.1615/jlongtermeffmedimplants.2013010238. PMID 25272207
- [Background] Slane J, Gietman B, Squire M. Antibiotic elution from acrylic bone cement loaded with high doses of tobramycin and vancomycin. J Orthop Res. 2018 Apr;36(4):1078-1085. doi: 10.1002/jor.23722. Epub 2017 Sep 20. PMID 28876459
- [Background] Anagnostakos K, Wilmes P, Schmitt E, Kelm J. Elution of gentamicin and vancomycin from polymethylmethacrylate beads and hip spacers in vivo. Acta Orthop. 2009 Apr;80(2):193-7. doi: 10.3109/17453670902884700. PMID 19404802